CLINICAL TRIAL: NCT05557747
Title: Cervicothoracic Junction Mobilization Versus Autogenic Muscle Energy Technique in Patients With Chronic Mechanical Neck Pain
Brief Title: Cervicothoracic Junction Mobilization Versus Muscle Energy Technique in Chronic Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hoda Ibrahim Abbas Mousa, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/003839
Record Dates: First submitted 2022-09-24; First posted 2022-09-28 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Chronic Mechanical Neck Pain
Keywords: chronic mechanical neck pain; cervicothoracic junction mobilization; autogenic muscle energy technique; cervicothoracic junction hypomobility

STUDY DESIGN:
Intervention Model Description: 1. mobilization and conventional physical therapy
  2. autogenic muscle Energy Technique and conventional physical therapy
  3. conventional physical therapy only
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A:cervicothoracic junction mobilization (Experimental): Group A: patients will receive cervicothoracic junction mobilization and conventional physical therapy program for 3 sessions/week over 4 weeks periods
  Interventions: Other: cervicothoracic junction mobilization in form of Maitland mobilization; Other: conventional physical therapy
- Group B:autogenic muscle Energy Technique (Experimental): Group B: will receive autogenic muscle Energy Technique and conventional physical therapy program for 3 sessions/week over 4 weeks periods.
  Interventions: Other: autogenic muscle Energy Technique; Other: conventional physical therapy
- Group C:conventional physical therapy (Active Comparator): Group C: will receive conventional physical therapy only in form of: (superficial heat using hot pack for 10 minutes , Isometric Neck Exercises and Dynamic Neck Exercises)) for 3 sessions/week over 4 weeks periods.
  Interventions: Other: conventional physical therapy

INTERVENTIONS:
Other: cervicothoracic junction mobilization in form of Maitland mobilization — Group A: will receive cervicothoracic junction mobilization mobilization in form of Maitland mobilization to the C7-T1 level, according to their primary movement restriction (for flexion-extension restriction- central PA glide, for rotation restrictions (unilateral PA glide) for 3 sessions/week over 4 weeks periods.
  Arms: Group A:cervicothoracic junction mobilization
Other: autogenic muscle Energy Technique — the technique will applied to neck muscles that are prone to get short including anterior, middle and posterior Scaleni, Sternocleidomastoid, Levator Scapulae and upper fibers of the Trapezius muscle.
  The AI MET group will given 3-5 repetitions of post isometric relaxation (PIR) (30-50% isometric contraction of the muscle to be stretched for 7-10 seconds, followed by rest period of 5 seconds and then a stretch of 10-60 seconds hold
  Arms: Group B:autogenic muscle Energy Technique
Other: conventional physical therapy — conventional physical therapy only in form of: (superficial heat using hot pack for 10 minutes , Isometric Neck Exercises and Dynamic Neck Exercises)) for 3 sessions/week over 4 weeks periods

SUMMARY:
This study will be conducted to identify the difference between the effect of of cervicothoracic junction mobilization and autogenic Muscle Energy Technique. on neck pain, cervical range of motion, cervical proprioception and neck disability in mechanical neck pain patients with cervicothoracic junction hypomobility.

ELIGIBILITY:
Inclusion criteria:

* Patients with a primary complaint of chronic neck pain (assessed by VAS )for more than 3 months
* Subjects with pain provocation and reduced mobility at the CT junction segment (assessed by passive accessory intervertebral movements (PAIVMs) and reduced mobility at cervical spine (assessed by CROM device.
* patients with age range from 18 to 45 years old.
* patients with body mass index less than 30 kg/m2.
* Exclusion Criteria:
* previous spine surgery
* pregnancy.
* Diabetic patients
* Hypertensive patients
* Patients were excluded if neck pain was associated with cervical radiculopathy
* whiplash injuries or severe headaches
* cervical spine fracture
* vertebro-basilar insufficiency.
* red flags suggesting of cancer, infection, vascular insufficiency
* Rheumatologic condition as mild systemic lupus erythematosus, poly-articular osteoarthritis, rheumatoid arthritis and advanced cervical spine degenerative diseases.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
change in neck pain | Evaluation Will be performed prior to the first treatment session; as a baseline measure, and at last treatment session(after 4 weeks) as a post-treatment measure
  change in neck pain will be measured by Visual analog scale for the 3 groups pre- and post treatment

SECONDARY OUTCOMES:
cervical ROM and cervical prorprioception | Evaluation Will be performed prior to the first treatment session; as a baseline measure, and at last treatment session(after 4 weeks) as a post-treatment measure
  cervical ROM and cervical prorprioception will be measured by cervical ROM device pre treatment and post treatment

CONTACTS AND LOCATIONS:
Locations (1):
- FACULTY OF PHYSICAL THERAPY, cairo university, Giza, Egypt